CLINICAL TRIAL: NCT03944382
Title: What Are the Effects of Fibrinogen Concentrate Administration on Biological Parameters
Acronym: Fibri_retro
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Fibri_retro
Record Dates: First submitted 2019-02-25; First posted 2019-05-09 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the fibrinogen concentrate are given since 50 years with the dose of 2g for a afibrinogenemia. But this dose has been fixed 40 years ago and from now nobody discuss this quantity. Through this retrospective study the investigators tried to explore the evolution of blood test after a prescription of fibrinogen concentrate

DETAILED DESCRIPTION:
the fibrinogen concentrate are given since 50 years with the dose of 2g for a afibrinogenemia. But this dose has been fixed 40 years ago and from now nobody discuss this quantity. Through this retrospective study the investigators tried to explore the evolution of blood test after a prescription of fibrinogen concentrate.

ELIGIBILITY:
Inclusion Criteria:

* all patient who received fibrinogen concentrate

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient who received fibrinogen concentrate
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Evolution of fibrinogen | one day
  Fibrinogen was measured before and after a fibrinogen factor transfusion. It will be used to calculate the delta (after - before) and mesure the efficiency of a transfusion
Evolution of FIBTEM A5® | one day
  FIBTEM A5® was measured before and after a fibrinogen factor transfusion. It will be used to calculate the delta (after - before) and mesure the efficiency of a transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DURANTEAU, Trainee, Principal Investigator — Erasme UH

IPD SHARING:
Plan to Share IPD: Undecided